CLINICAL TRIAL: NCT02373956
Title: Evaluation of the Efficacy and Tolerance of Honey-impregnated Dressings Versus Non-impregnated Dressings in the Local Management of Pressure Ulcers: A Randomized Single-blind Trial
Brief Title: Efficacy and Tolerance of Honey-impregnated Dressings in the Local Management of Pressure Ulcers
Acronym: MeliCare
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties to include
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: MELIPHARM SAS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LOCAL/2014/JPL-01; 2014-A01407-40 (Other: RCB number)
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MELECTIS G (Experimental): In addition to usual care as described for the other arm, patients randomized to this arm will have MELECTIS G added to their wound dressing according to the manufacturer's instructions.
  Intervention: Usual care Intervention: MELECTIS G
  Interventions: Device: MELECTIS G
- Usual care (Active Comparator): Patients randomized to this are will receive usual care according the current procedures at the Nîmes University Hospital (ICMD010 concerning pressure sore care and SCMD002 concerning referenced anti-pressure sore dressings).
  Intervention: Usual care
  Interventions: Device: MELECTIS G; Procedure: Usual care

INTERVENTIONS:
Device: MELECTIS G — The experimental medical device (MELECTIS G) is an association of selected honey and pharmaceutical grade hyaluronic acid.
Procedure: Usual care — Patients will receive usual care according to the current procedures at the Nîmes University Hospital (ICMD010 concerning pressure sore care and SCMD002 concerning referenced anti-pressure sore dressings).
  Arms: Usual care

SUMMARY:
The main objective of this study is to document the effectiveness of a honey-based medical device (Hyalumel) in the management of pressure ulcers. The effectiveness of the medical device will be judged according to the evolution of the surface of the wound at the end of 12 weeks of treatment.

DETAILED DESCRIPTION:
The secondary objectives of this study are to compare the following items between the two arms of the study:

A. The evolution of skin microbiota in the wound B. The evolution of the surface and the depth of the wound during follow-up C. The healing process D. Patient and caretaker acceptability

ELIGIBILITY:
Inclusion Criteria:

* Information provided on the implementation of the study, its objectives, constraints and patient rights
* The patient, or his/her legal guardian, must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 12 weeks of follow-up
* Presence of one or more pressure ulcers at stages 2, 3 or 4 according to the European Pressure Ulcer Advisory Panel - National Pressure Ulcer Advisory Panel (EPUAP-NPUAP) classification
* Wound whose surface is between 1 cm^2 and 15 cm^2
* Wound present for more than 6 weeks
* Patient whose wound requires a modern dressing (that is to say, a bandage that is neither tulle nor gauze) without bactericidal agents or antibiotics
* No antibiotics for at least 7 days prior to inclusion (after inclusion, the patient can be treated with antibiotics if necessary, regardless of the indications)

Exclusion Criteria:

* Patient participating in or having participated in another interventional study in the previous 3 months or currently in a patient exclusion period determined by a previous study.
* Patient under judicial protection
* Failure to correctly inform the patient or his/her legal representative
* Patient (or his/her legal guardian) refusal to sign the consent
* The patient is pregnant, parturient, or breastfeeding
* Contraindications (or incompatible combination therapy) for a necessary treatment in this study
* Patient with an allergy to honey or propolis
* The patient's general condition suggests study exclusion before twelve weeks of follow-up
* Antibiotics received within 7 days prior to inclusion
* Active neoplastic lesion treated with radiation or chemotherapy
* Immunosuppressive therapy or other treatment which, in the judgment of the investigator, may interfere with the healing process
* Surgery planned within twelve weeks of inclusion
* Stage 1 wound according to the EPUAP-NPUAP classification
* Amputation wound
* Wound related to a surgical treatment or for which an act of revascularization is envisaged within twelve weeks of inclusion
* Malignant wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Change in wound surface area according to the Gilman formula | Week 12
  According to the Gilman formula

SECONDARY OUTCOMES:
Change in wound surface area according to the Gilman formula | Week 1
  According to the Gilman formula
Change in wound surface area according to the Gilman formula | Week 2
  According to the Gilman formula
Change in wound surface area according to the Gilman formula | Week 4
  According to the Gilman formula
Change in wound surface area according to the Gilman formula | Week 8
  According to the Gilman formula
Change in wound surface area according to the Gilman formula | Week 12
  According to the Gilman formula
Change in wound surface area according to the Gilman formula | At treatment stopping if appropriate (before week 12)
  According to the Gilman formula
Relative variation (%) in wound surface area | Week 1
Relative variation (%) in wound surface area | Week 2
Relative variation (%) in wound surface area | Week 4
Relative variation (%) in wound surface area | Week 8
Relative variation (%) in wound surface area | Week 12
Relative variation (%) in wound surface area | At treatment stopping if appropriate (before week 12)
Relative variation (%) in wound depth | Week 1
Relative variation (%) in wound depth | Week 2
Relative variation (%) in wound depth | Week 4
Relative variation (%) in wound depth | Week 8
Relative variation (%) in wound depth | Week 12
Relative variation (%) in wound depth | At treatment stopping if appropriate (before week 12)
Has the wound surface area reduced by at least 40%? yes/no | Week 2
Has the wound surface area reduced by at least 40%? yes/no | Week 4
Has the wound surface area reduced by at least 40%? yes/no | Week 8
Has the wound surface area reduced by at least 40%? yes/no | Week 12
Has the wound surface area reduced by at least 40%? yes/no | At treatment stopping if appropriate (before week 12)
Number of bacteria species present in the wound | Baseline (Day 0)
Number of bacteria species present in the wound | Day 14
Number of bacteria species present in the wound | Day 84
Diversity (Shannon's H) of bacteria species present in the wound | Baseline (Day 0)
Diversity (Shannon's H) of bacteria species present in the wound | Day 14
Diversity (Shannon's H) of bacteria species present in the wound | Day 84
Number of bacteria functional groups present in the wound | Baseline (Day 0)
  Functional groups: commensal, pathogenic, weak pathogenic potential
Number of bacteria functional groups present in the wound | Day 14
  Functional groups: commensal, pathogenic, weak pathogenic potential
Number of bacteria functional groups present in the wound | Day 84
  Functional groups: commensal, pathogenic, weak pathogenic potential
Diversity (Shannon's H) of bacteria functional groups present in the wound | Baseline (Day 0)
  Functional groups: commensal, pathogenic, weak pathogenic potential
Diversity (Shannon's H) of bacteria functional groups present in the wound | Day 14
  Functional groups: commensal, pathogenic, weak pathogenic potential
Diversity (Shannon's H) of bacteria functional groups present in the wound | Day 84
  Functional groups: commensal, pathogenic, weak pathogenic potential
The number of multiresistant bacteria species present in the wound | Baseline (Day 0)
The number of multiresistant bacteria species present in the wound | Day 14
The number of multiresistant bacteria species present in the wound | Day 84
the ratio of the number of commensal over the total number of bacteria species present in the wound | Baseline (Day 0)
the ratio of the number of commensal over the total number of bacteria species present in the wound | Day 14
the ratio of the number of commensal over the total number of bacteria species present in the wound | Day 84
the ratio of the number of commensal or weakly virulent over the total number of bacteria species present in the wound | Baseline (Day 0)
the ratio of the number of commensal or weakly virulent over the total number of bacteria species present in the wound | Day 14
the ratio of the number of commensal or weakly virulent over the total number of bacteria species present in the wound | Day 84
Wound healing speed (change in cm^2 of surface area per week) | 12 weeks (or maximum time span if total healing occurs before 12 weeks)
Is the wound completely healed? yes/no | Week 12
The time to healing (days) | Week 12
Appearance of the pressure ulcer | Baseline (Day 0)
  Appearance of the pressure ulcer: burgeoning, fibrinous, necrotic, blistering or de-epidermisation, exudative, bad odor
Appearance of the pressure ulcer | Week 1
  Appearance of the pressure ulcer: burgeoning, fibrinous, necrotic, blistering or de-epidermisation, exudative, bad odor
Appearance of the pressure ulcer | Week 2
  Appearance of the pressure ulcer: burgeoning, fibrinous, necrotic, blistering or de-epidermisation, exudative, bad odor
Appearance of the pressure ulcer | Week 4
  Appearance of the pressure ulcer: burgeoning, fibrinous, necrotic, blistering or de-epidermisation, exudative, bad odor
Appearance of the pressure ulcer | Week 8
  Appearance of the pressure ulcer: burgeoning, fibrinous, necrotic, blistering or de-epidermisation, exudative, bad odor
Appearance of the pressure ulcer | Week 12
  Appearance of the pressure ulcer: burgeoning, fibrinous, necrotic, blistering or de-epidermisation, exudative, bad odor
Appearance of the pressure ulcer | At treatment stopping if appropriate (before week 12)
  Appearance of the pressure ulcer: burgeoning, fibrinous, necrotic, blistering or de-epidermisation, exudative, bad odor
Presence/absence of adverse events | Week 1
Presence/absence of adverse events | Week 2
Presence/absence of adverse events | Week 4
Presence/absence of adverse events | Week 8
Presence/absence of adverse events | Week 12
Presence/absence of adverse events | At treatment stopping if appropriate (before week 12)
Algo plus scale | Baseline (Day 0)
Algo plus scale | Week 1
Algo plus scale | Week 2
Algo plus scale | Week 4
Algo plus scale | Week 8
Algo plus scale | Week 12
Algo plus scale | At treatment stopping if appropriate (before week 12)
Acceptability of the dressing by the medical staff | Week 1
  Acceptability of the dressing by the medical staff in relation to each of the following:
  * Overall satisfaction
  * Easy installation
  * Ease of removal
  * conformability of the dressing to the wound
  * Pain at dressing change
  * Adhesion of dressing to the wound
Acceptability of the dressing by the medical staff | Week 2
  Acceptability of the dressing by the medical staff in relation to each of the following:
  * Overall satisfaction
  * Easy installation
  * Ease of removal
  * conformability of the dressing to the wound
  * Pain at dressing change
  * Adhesion of dressing to the wound
Acceptability of the dressing by the medical staff | Week 4
  Acceptability of the dressing by the medical staff in relation to each of the following:
  * Overall satisfaction
  * Easy installation
  * Ease of removal
  * conformability of the dressing to the wound
  * Pain at dressing change
  * Adhesion of dressing to the wound
Acceptability of the dressing by the medical staff | Week 8
  Acceptability of the dressing by the medical staff in relation to each of the following:
  * Overall satisfaction
  * Easy installation
  * Ease of removal
  * conformability of the dressing to the wound
  * Pain at dressing change
  * Adhesion of dressing to the wound
Acceptability of the dressing by the medical staff | Week 12
  Acceptability of the dressing by the medical staff in relation to each of the following:
  * Overall satisfaction
  * Easy installation
  * Ease of removal
  * conformability of the dressing to the wound
  * Pain at dressing change
  * Adhesion of dressing to the wound
Acceptability of the dressing by the medical staff | At treatment stopping if appropriate (before week 12)
  Acceptability of the dressing by the medical staff in relation to each of the following:
  * Overall satisfaction
  * Easy installation
  * Ease of removal
  * conformability of the dressing to the wound
  * Pain at dressing change
  * Adhesion of dressing to the wound

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Lavigne, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - Centre Mutualiste Neurologique Propara, Montpellier
  - CHRU de Nîmes - Centre de Gérontologie de Serre Cavalier, Nîmes
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes